CLINICAL TRIAL: NCT07143487
Title: Evaluation of Provider vs. Patient Mediated Cascade Genetic Testing of First-Degree Relatives of Patients With Newly Diagnosed Colorectal Cancer
Brief Title: Family Communications After Genetic Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: A212101
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Colon Adenocarcinoma; Colorectal Adenocarcinoma; Rectal Adenocarcinoma; Stage I Colon Cancer AJCC v8; Stage I Colorectal Cancer AJCC v8; Stage I Rectal Cancer AJCC v8; Stage II Colon Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage II Rectal Cancer AJCC v8; Stage III Colon Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IV Colon Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Rectal Cancer AJCC v8
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Step 1 (biospecimen collection, genetic testing) (Experimental): Probands undergo collection of blood samples and genetic testing on study.
  Interventions: Procedure: Biospecimen Collection; Other: Genetic Testing
- Step 2, Arm A (proband-mediated) (Active Comparator): FDRs receive proband-mediated communication about the proband's genetic testing results.
  Interventions: Other: Communication Intervention; Other: Survey Administration
- Step 2, Arm B (provider-mediated) (Experimental): FDRs receive provider-mediated communication about the proband's genetic testing results.
  Interventions: Other: Communication Intervention; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Arms: Step 1 (biospecimen collection, genetic testing)
Other: Genetic Testing — Undergo genetic testing
  Arms: Step 1 (biospecimen collection, genetic testing)
Other: Communication Intervention — Receive proband-mediated communication
  Arms: Step 2, Arm A (proband-mediated); Step 2, Arm B (provider-mediated)
Other: Survey Administration — Ancillary studies
  Arms: Step 2, Arm A (proband-mediated); Step 2, Arm B (provider-mediated)

SUMMARY:
This clinical trial compares patient (proband)-mediated communication to provider-mediated communication for improving genetic testing in first-degree relatives of patients with newly diagnosed colorectal cancer. It is estimated that 30% of cases of colorectal cancer have a genetic basis and about 15% of these patients have a disease-causing (pathogenic) inherited (germline) variant in a cancer susceptibility gene. Most individuals carrying a pathogenic germline variant are unaware of their cancer risk and may not meet guidelines for genetic testing. Identifying pathogenic germline variants or hereditary cancer syndromes in cancer patients has important implications for their at-risk relatives who may not know that they are at high risk for cancer. The burden of communicating this risk to first-degree relatives often falls on the patients, who may lack sufficient knowledge to correctly share and explain their genetic test results. Receiving provider-mediated communication of genetic testing results may be more effective at communicating genetic risk to first-degree relatives than the usual practice of proband-mediated communication.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the proportion of first-degree relatives (FDRs) of probands with Lynch Syndrome who undergo germline testing in the provider-mediated arm (Arm B) versus the proband-mediated (Arm A) at 6 months.

II. To compare the proportion of FDRs of proband with a non-Lynch pathogenic germline variant who undergo germline testing in the provider-mediated arm (Arm B) versus the proband-mediated arm (Arm A) at 6 months.

SECONDARY OBJECTIVE:

I. To compare the proportion of FDRs with a pathogenic germline variant (PGV) who underwent disease prevention efforts at 12 months between the provider-mediated arm (Arm B) and the proband-mediated cascade testing arm (Arm A).

EXPLORATORY OBJECTIVES:

I. To assess differences in percentages of cascade genetic testing within the following proband subgroups: race/ethnicity (non-Hispanic whites; other race/ethnicities), sex (females; males), age (>= 50; < 50), tumor location (colon; rectal), tumor stage (stage I-II; stage III-IV), geographic location (urban; rural), and receipt of medical care in an academic versus (vs.) community setting.

III. To determine the prevalence and spectrum of pathogenic germline variants in cancer susceptibility genes by analysis of results of upfront germline testing in a multi-site cancer cooperative group study population with newly diagnosed CRC.

IV. Assess the pattern of accrual of demographic patient subgroups including racial/ethnic minority and rural individuals at the initial 50% of accrual enrolled and at the end of the trial.

V. To compare disease-free survival (DFS) of the proband at 3 years between the direct-contact arm (Arm B) and the proband-directed cascade testing arm (Arm A).

V. To evaluate the completion rate of a Social Determinants of Health questionnaire with patient directed questions .

OUTLINE:

STEP 1: Patients (probands) undergo collection of blood samples and genetic testing on study.

STEP 2: Probands with pathogenic or likely pathogenic germline variants and their FDRs are randomized to 1 of 2 arms.

ARM A: FDRs receive proband-mediated communication about the proband's genetic testing results.

ARM B: FDRs receive provider-mediated communication about the proband's genetic testing results.

Probands are followed for up to 3 years and FDRs are followed for up to 1 year

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 PROBANDS: Age >= 18 years
* STEP 1 PROBANDS: Patients with a newly diagnosed (within 3 months of registration), primary colorectal adenocarcinoma, stage I to IV

  * Histologically proven stage I to IV colon or rectal adenocarcinoma (any T or N, M+). Tumors deemed to originate in the colon can extend into/involve the small bowel (e.g., those at the ileocecal valve). Tumors will be regarded as originating in the colon if the entire tumor is in the colon. In the case of rectal involvement, the cancer will be considered a rectal primary
  * Patients with more than one primary colon adenocarcinoma are eligible
* STEP 1 PROBANDS: No patients with stage 0 or in-situ colorectal cancer
* STEP 1 PROBANDS: Patients who have had prior malignancies are eligible, including non-invasive cancers
* STEP 1 PROBANDS: Patients with synchronous second malignancies are eligible
* STEP 1 PROBANDS: Have not received germline testing in the 2 years prior to enrollment or known hereditary colon cancer syndromes
* STEP 1 PROBANDS: Patients must have at least 2 living FDRs who meet the eligibility criteria, with whom the patient is willing to share their cancer diagnosis
* STEP 1 PROBANDS: In order to complete the mandatory patient-completed measures and view the video and receive genetic education and counseling, participants must be able to speak and read English or Spanish
* STEP 1 PROBANDS: No known diagnosis of dementia or cognitive impairment. Persons with impaired decision-making capacity are ineligible as they need to be able to understand genetic test results, its implications for the patient and family, and explain genetic test results to their family members

  * No persons with a known psychiatric or documented developmental disorder that affects cognitive or emotional functions to the extent that the capacity for judgment and reason is significantly diminished, such that they cannot participate based on the judgment of the treating physician
* STEP 2 PROBANDS: Probands positive for a pathogenic germline variant (PGV) in a cancer susceptibility gene
* FDRs: Age >= 18 years
* FDRs: Have not previously received germline genetic testing or known hereditary colon cancer syndromes
* FDRs: FDRs must reside within the United States, as genetic testing from LabCorp is only available to United States (U.S.) residents
* FDRs: In order to complete the mandatory patient-completed measures, participants must be able to speak and read English or Spanish

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4186 (Estimated)
Dates: Start 2025-11-05 (Estimated); Primary Completion 2029-11-05 (Estimated); Study Completion 2032-11-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible first-degree relatives (FDRs) of the affected proband who underwent genetic testing | Within 6 months of proband randomization
  This is a binary outcome. To test for a between-arm difference in the proportion of eligible FDRs receiving genetic testing, the primary analysis will apply a mixed-effects logistic regression model to account for between-family variability or equivalently the within family correlation. The mixed-effects logistic regression model will be applied separately within the subset of families who are associated with a proband who has Lynch syndrome (LS), and within the subset of families who are associated with a proband who harbors non-LS pathogenic germline variants (PGVs).

SECONDARY OUTCOMES:
Proportion of eligible FDRs with a PGV undergoing disease prevention efforts | Within 12 months of proband randomization
  Binary outcome indicating whether an eligible FDR with a PGV who underwent disease prevention efforts at 12 months between the provider-mediated arm (Arm B) and the proband-mediated cascade testing arm (Arm A).

OTHER OUTCOMES:
Proportion of eligible FDRs of the affected proband who underwent genetic testing | Within 6 months of proband randomization
  Will repeat LS and non-LS analyses according to pre-defined proband sub-groups (Non-Hispanic White vs. other races/ethnicities; female vs. male; age >= 50 vs. < 50; urban vs. rural; academic setting vs. community setting). It is clinically important to quantify the effect of the provider-mediated direct-contact approach within these subgroups and the degree of imprecision as measured by the corresponding confidence interval. Thus, we will report the odds ratio and descriptive 95% confidence interval.
Degree to which the somatic tumor profiling identifies a germline event | up to 3 years
  Will estimate the proportion of cases where the germline mutation is detected by somatic next generation sequencing testing of the tumor. The corresponding lower bound of the one-sided 90% interval will be calculated for the true but unknown proportion.
Spectrum and prevalence of PGVs in cancer susceptibility genes | Up to 3 years
  For each, descriptive statistics will include the frequency and percentage as well as the standard error.
Disease-free survival (DFS) of probands | From the date the patient is randomized on study for first documentation of primary tumor recurrence/relapse or death, assessed up to 3 years
  : DFS will be compared between direct-contact arm and proband-directed cascade testing arm. DFS percentages, standard errors, and the intervention effect comparison will be obtained from the Kaplan-Meier method, Greenwood's formula, and log-rank tests, respectively. Cox proportional hazards regression models will be used to estimate relative risks and 95% confidence intervals for the intervention comparison.
Accrual patterns | up to 3 years
  Summary of participant accrual over time, including recruitment rates by site and arm.

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Sinicrope, Study Chair — Alliance for Clinical Trials in Oncology

IPD SHARING:
Plan to Share IPD: Undecided